CLINICAL TRIAL: NCT04971096
Title: Relationship Between Gut Microbiome, Probiotics, and Mild Cognitive Impairment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult to include the patient.
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: Bened Biomedical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shu-I Wu, Senior Attending Physician, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20CT060be
Record Dates: First submitted 2021-06-25; First posted 2021-07-21 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment (MCI)
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participates in three groups, 60 patients in each group. One group of patients will be given PS23, one will be given heat-treated PS23 and the other one will be given placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a double blind randomized control study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PS23 (Experimental): The PS23 belongs to Lactobacillus paracasei group, 2 caps daily use.
  Interventions: Dietary Supplement: PS23 live
- heat-treated PS23 (Experimental): PS23 heat-treated, 2 caps daily use.
  Interventions: Dietary Supplement: PS23 heat-treated
- placebo (Placebo Comparator): The placebo capsule contains microcrystalline cellulose, 2 caps daily use.
  Interventions: Dietary Supplement: Placebo
- Healthy Control (No Intervention): No intervention

INTERVENTIONS:
Dietary Supplement: PS23 live — PS23 belongs to Lactobacillus paracasei group.Probiotic capsules contain 30 billion CFU (colony forming units) of PS23
  Arms: PS23
Dietary Supplement: PS23 heat-treated — The PS23 heat-treated probiotic capsule contain 30 billion of PS23 cells.
  Arms: heat-treated PS23
Dietary Supplement: Placebo — The placebo capsule contains microcrystalline cellulose.
  Arms: placebo

SUMMARY:
This study is to evaluate whether the consumption of probiotics can improve the symptoms of patients with mild cognitive impairment; also evaluate the effects of probiotics on patients' blood, oxidation and stress related indicators.

DETAILED DESCRIPTION:
Mild cognitive impairment (MCI) is the stage between the expected cognitive decline of normal aging and the more serious decline of dementia. It can involve problems with memory, language, thinking and judgment that are greater than normal age-related changes. Probiotics are regarded as active microorganisms. When consumed in sufficient amounts, participants can regulate intestinal flora, intestinal permeability, inflammation and antioxidant reactions in the body, and may produce host health, including delaying disease and regulating metabolic disease progression and prevent complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who is suffering from Mild Cognitive Impairment.
2. Clinical Dementia Rating (CDR) 0.5.
3. Age 40-80 and willing to sign the Informed Consent.
4. Education level is above the junior high school level.
5. Healthy control who is eligible judged by PI.

Exclusion Criteria:

1. Patients on antibiotics within the preceding one month.
2. Patients using of other probiotic products (sachet, capsule or tablet) within the preceding two weeks.
3. Have undergone surgery of liver, bladder, or gastrointestinal tract.
4. Have current or history of inflammatory bowel disease.
5. Have history of cancer.
6. Known allergy to probiotics.
7. Dementia (MMSE ≤ 23).
8. Cognitive Impairment caused by head injury.
9. History of cerebral apocalypse.
10. Other possible diseases may cause cognitive impairment, such as: Parkinson's disease, cervical mass, hydrocephalus or epilepsy.
11. Severely depressed patients (sick person health questionnaire-9 (PHQ-9) ≥ 20).
12. Severe anxiety patients (Generalized Anxiety Dosorder 7-Item (GAD-7) ≧ 15).
13. Undergoing medication treatment for acute illness, Organic psychosis or diagnosed as psychiatric illness within 3 months or poor control of chronic psychiatric illness.
14. Undergoing parenteral nutrition.
15. Not eligible judged by PI.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination, MMSE (end point scare-baseline score)/ Baseline score*100% ≥ 12% | From Baseline to 12 Weeks Assessed
  The Mini-Mental State Exam (MMSE) is a widely used test of cognitive function, The maximum MMSE score is 30 points. A score of 20 to 24 suggests mild dementia, 13 to 20 suggests moderate dementia among the elderly; it includes tests of orientation, attention, memory, language and visual-spatial skills.
Wechsler Memory Scale-III, WMS-III (end point scare-baseline score)/ Baseline score*100% ≥ 12% | From Baseline to 12 Weeks Assessed
  The WMS-III has most representative standardization databases to assess memory and make optimal clinical recommendations. The 11 subtests that comprise the index scores average 60 min, ranging from 45 to 75 min, to administer. The time needed to administer the 13 subtests required to generate all of the summary and index scores is 80 min, with a range of 65 to 95 min.

SECONDARY OUTCOMES:
Change in Cognitive Abilities Screening Instrument, CASI | From Baseline to 12 Weeks Assessed
  The Cognitive Abilities Screening Instrument (CASI) has a score range of 0 to 100 and provides quantitative assessment on attention, concentration, orientation, short-term memory, long-term memory, language abilities, visual construction, list-generating fluency, abstraction, and judgment, higher scores mean a better outcome.
Change in Clinical Dementia Rating (CDR) | From Baseline to 12 Weeks Assessed
  The CDR is a global summary measure designed to identify the overall severity of dementia. Six different content areas are rated individually (memory, orientation, judgement and problem solving, community affairs, home and hobbies, and personal care). CDR is calculated on the basis of testing six different cognitive and behavioral domains such as memory, orientation, judgment and problem solving, community affairs, home and hobbies performance, and personal care. The CDR is based on a scale of 0-3: no dementia (CDR = 0), questionable dementia (CDR = 0.5), MCI (CDR = 1), moderate cognitive impairment (CDR = 2), and severe cognitive impairment (CDR = 3).
Change in Insomnia Severity Index, ISI | From Baseline to 12 Weeks Assessed
  The ISI is a rating tool used to gauge of sleeping. Higher values represent a worse outcome. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Change in Geriatric Depression Scale, GDS | From Baseline to 12 Weeks Assessed
  The Geriatric Depression Scale (GDS) is a self-report measure of depression in older adults. Users respond in a "Yes/No" format. The GDS was originally developed as a 30-item instrument. Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
Change in Hamilton Anxiety Scale, HAM-A | From Baseline to 12 Weeks Assessed
  The HAM-A was one of the first rating scales developed to measure the severity of anxiety symptoms, and is still widely used today in both clinical and research settings. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Change in The Quality of Life, Enjoyment, and Satisfaction Questionnaire-16, QLESQ-16 | From Baseline to 12 Weeks Assessed
  The Quality of Life, Enjoyment, and Satisfaction Questionnaire-16 is a valid, reliable self-report instrument for assessing quality of life. The minimum raw score on the Q-LES-Q-16 is 14, and the maximum score is 70, higher scores mean a better outcome.
Change in Visual Analogue Scale for GI symptoms (VAS-GI) | From Baseline to 12 Weeks Assessed
  Visual Analogue Scale for GI symptoms, VAS-GI (visual analogue scale, VAS 0-10) was designed to measure the response of symptoms and well-being in patients after taking PS23, total score is 0-100, higher scores mean a worse outcome.
Change in Color Trails Test (CTT) | From Baseline to 12 Weeks Assessed
  Color Trails Test (CTT) is developed to be free from the influence of language and cultural bias, the CTT assesses sustained attention in adults.
Change in levels of exploratory blood-based biomarkers for inflammatory and/or oxidative stress changes | From Baseline to 12 Weeks Assessed
  Blood-based biomarkers (e.g. IL-6, TNF-α, GDF-15, Adiponectin, EGF, BDNF, MDA, Nitric oxide (NO) , GSH, TAC, Ghrelin, Cystatin C , Hs-CRP, HbA1c, Glucose (AC), Triglycerides (TG), LDL, HDL , Insulin, miRNA and total cholesterol )
Change in Gut microbiome | From Baseline to 12 Weeks Assessed
  The gut microbiome plays important roles in both the maintenance of health and the pathogenesis of disease. Stool will be examined before and after probiotics.
Change in WAIS-IV | From Baseline to 12 Weeks Assessed
  WAIS-IV is composed of 10 core subtests and five supplemental subtests, with the 10 core subtests yielding scaled scores that sum to derive the Full Scale IQ. With the WAIS-IV, the verbal/performance IQ scores from previous versions were removed and replaced by the index scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan